CLINICAL TRIAL: NCT00202176
Title: The Effects of Bronchodilators on Exertional Dyspnea and Exercise Performance in Mild Chronic Obstructive Pulmonary Disease (COPD) Patients and Healthy Elderly Subjects.
Brief Title: Effects of Bronchodilators in Mild Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Dr. Denis O'Donnell, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DMED-833-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic; Obstructive; Pulmonary; Disease; COPD; Atrovent; Ipratropium; Bromide; Exercise; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Disease; Motor Activity; Dyspnea | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ipratropium Bromide
  Interventions: Drug: Ipratropium Bromide
- 2 (Placebo Comparator): Saline Solution (0.9% NaCl)
  Interventions: Drug: Ipratropium Bromide

INTERVENTIONS:
Drug: Ipratropium Bromide — Nebulized Ipratropium Bromide (4 mL) or saline solution (0.9% NaCl) (4mL) will be administered to subjects once only.
  Other Names: Atrovent

SUMMARY:
In people with mild COPD, the ability to exhale air from the lungs is partly limited because of narrowing and collapse of the airways. This results in the trapping of air within the lungs and over-distention of the lungs and chest (lung hyperinflation).

Breathing at high lung volumes (hyperinflation) is an important cause of breathing discomfort (dyspnea) in people with COPD. Bronchodilators help to relax muscles in the airways or breathing tubes. Bronchodilators are often prescribed if a cough occurs with airway narrowing as this medication can reduce coughing, wheezing and shortness of breath. Bronchodilators can be taken orally, through injection or through inhalation and begin to act almost immediately but with the effect only lasting 4-6 hours. The main purpose of this study is to examine the effects of inhaled bronchodilators on breathing discomfort and exercise endurance in patients with mild COPD.

DETAILED DESCRIPTION:
In people with mild COPD, the ability to exhale air from the lungs is partly limited because of narrowing and collapse of the airways. This results in the trapping of air within the lungs and over-distention of the lungs and chest - this is known as lung hyperinflation. We believe that breathing at high lung volumes (hyperinflation) is an important cause of breathing discomfort (dyspnea) in people with COPD. Bronchodilators help to relax muscles in the airways or breathing tubes. Bronchodilators are often prescribed if a cough occurs with airway narrowing; this medication can reduce coughing, wheezing and shortness of breath. Bronchodilators can be taken orally, through injection or through inhalation and begin to act almost immediately but with the effect only lasting 4-6 hours. The main purpose of this study is to examine the effects of inhaled bronchodilators on breathing discomfort and exercise endurance in patients with mild COPD.

Each subject will attend 4 visits to the laboratory. Visit 1 (screening visit) will involve a record of medical history, medications used, anthropometrics measurements, questionnaires, breathing tests, an incremental cycle exercise test and a constant-workload cycle exercise test. Visit 2 will involve breathing tests and a constant-workload cycle exercise test. Visits 3 and 4 will involve breathing tests and a constant-workload cycle exercise test after subjects have been randomized to either placebo or Atrovent. These visits will be done on separate days and subjects will receive the two above treatments in random order.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild COPD OR healthy control subjects
* 40-80 years old
* able to perform all study procedures
* Smoking history > 10 pack years (for mild COPD) or smoking history < 10 pack years (for healthy control subjects)

Exclusion Criteria:

* allergy to atrovent
* history of asthma, atopy or nasal polyps
* Oxygen desaturation < 80 % during exercise
* recent history of CAD (under a year) or any significant diseases that could contribute to dyspnea or exercise limitation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
endurance time | 2 hours post-study drug inhalation
dyspnea | 2 hours post-study drug inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Queen's University-Respiratory Investigation Unit
Locations (1):
- Respiratory Investigation Unit, Kingston, Ontario, Canada